CLINICAL TRIAL: NCT02979431
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Dose Ranging Study of ALX-0171 in Infants and Young Children Hospitalized for Respiratory Syncytial Virus Lower Respiratory Tract Infection
Brief Title: Dose Ranging Study of ALX-0171 in Infants Hospitalized for Respiratory Syncytial Virus Lower Respiratory Tract Infection
Acronym: Respire
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0171-C201; 2016-001651-49 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Syncytial Virus Lower Respiratory Tract Infection
Keywords: RSV, Lower Respiratory Tract Infection, pediattric patients
MeSH Terms: interventions — gontivimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ALX-0171 3.0 mg/kg (Experimental): Inhalation of ALX-0171 3.0 mg/kg once daily for 3 consecutive days
  Interventions: Biological: ALX-0171 3.0 mg/kg
- ALX-0171 6.0 mg/kg (Experimental): Inhalation of ALX-0171 6.0 mg/kg once daily for 3 consecutive days
  Interventions: Biological: ALX-0171 6.0 mg/kg
- ALX-0171 Dose 9.0mg/kg (Experimental): Inhalation of ALX-0171 9.0 mg/kg once daily for 3 consecutive days
  Interventions: Biological: ALX-0171 9.0 mg/kg
- Placebo (Placebo Comparator): Inhalation of Placebo once daily for 3 consecutive days
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ALX-0171 3.0 mg/kg
  Arms: ALX-0171 3.0 mg/kg
Biological: ALX-0171 6.0 mg/kg
  Arms: ALX-0171 6.0 mg/kg
Biological: ALX-0171 9.0 mg/kg
  Arms: ALX-0171 Dose 9.0mg/kg
Other: Placebo
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the anti-viral effect and safety of different doses of inhaled ALX-0171 in subjects hospitalized for Respiratory Syncytial Virus Lower Respiratory Tract Infection (RSV LRTI). The secondary objective is to evaluate the clinical activity, pharmacokinetic (PK) properties, pharmacodynamic (PD) effect and immunogenicity of different doses of inhaled ALX-0171.

DETAILED DESCRIPTION:
This was a Phase 2b, randomized, double-blind, placebo-controlled, international, multicenter dose-ranging study in infants and toddlers hospitalized for RSV LRTI. The study evaluated 3 dose levels of ALX-0171 in a sequential part (safety Cohorts 1-3) followed by a parallel part (Cohort 4).

An Independent Data Monitoring Committee (IDMC) was assigned to review study data and provide recommendations on proceeding to the next safety cohort and on which dose levels could be taken forward in the parallel part.

Three dose levels of ALX-0171 were evaluated:

* Dose 1: target dose of 3.0 mg/kg
* Dose 2: target dose of 6.0 mg/kg
* Dose 3: target dose of 9.0 mg/kg

The study drug was administered by inhalation once daily for 3 consecutive days along with standard of care treatment, which was determined by the Investigator (or his/her designee) according to institutional practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infant or young child aged 28 days to < 2 years with gestational age ≥ 33 weeks at screening.
2. Subject weighed between ≥ 3.0 kg and < 15.0 kg at screening.
3. Subject is otherwise healthy but was hospitalized for and clinically diagnosed with RSV LRTI (bronchiolitis or broncho-pneumonia), i.e., showing typical clinical signs and symptoms such as tachypnea, wheezing, cough, crackles, use of accessory muscles and/or nasal flaring.
4. Subject had a positive RSV diagnostic test at screening.
5. Subject was expected to have to stay in the hospital for at least 24 hours (according to the Investigator's judgment at screening).
6. Symptoms were likely related to RSV infection (i.e., the symptoms present needed to be probably linked to the current RSV infection according to Investigator's judgment) had appeared within 4 days of screening and were not yet improving at screening and randomization.
7. Subject fulfilled at least 2 of the following RSV disease severity criteria at screening and randomization:

   * Inadequate oral feeding that required feeding support (i.e., nasogastric tube or intravenous [i.v.] line)
   * Inadequate oxygen saturation defined as:

     * Oxygen saturation (peripheral capillary oxygen saturation [SpO2]) ≤ 92% on room air or
     * Requiring oxygen supplementation to maintain oxygen saturation > 90% with documented pre-supplementation value ≤ 92%
   * Signs of respiratory distress defined as:

     * Respiratory rate ≥ 50 per minute in infants up to 12 months of age, and ≥ 40 per minute in children above 12 months and/or
     * Moderate or marked respiratory muscle retractions
8. Normal psychomotor development.

Exclusion Criteria:

1. Subject was known to have significant comorbidities including:

   * Genetic disorders (e.g., trisomy 21, cystic fibrosis),
   * Hemodynamically significant congenital heart disease (e.g., needing corrective therapy or inotropic support),
   * Bronchopulmonary dysplasia,
   * Any hereditary or acquired metabolic (bone) diseases,
   * Hematologic or other malignancy.
2. Subject was known to be human immunodeficiency virus (HIV)-positive. If the subject was < 6 months of age, a known HIV-positivity of the mother was also exclusionary.
3. Subject was known to be immunocompromised.
4. Subject had or was suspected to have an active, clinically relevant concurrent infection (e.g., bacterial pneumonia, urinary tract infection). Concurrent acute otitis media was not exclusionary.
5. Subject had significant oral and/or maxillofacial malformations that would prevent proper positioning of the face mask.
6. Subject received invasive mechanical ventilation or non-invasive respiratory support (i.e., continuous or bilevel positive airway pressure) in the 4 weeks prior to screening.
7. During the admission, the subject was initially hospitalized in an intensive care unit (ICU) setting and/or had received invasive mechanical ventilation or non-invasive respiratory support (i.e., continuous or bilevel positive airway pressure).
8. Subject was critically ill and/or was expected to require invasive mechanical ventilation, non invasive respiratory support (i.e., continuous or bilevel positive airway pressure), or High Flow oxygen therapy (HFOT) at levels not enabling nebulization therapy according to the Investigator's judgment. High Flow oxygen, with a maximum flow of 2 L/kg/min, was permitted under the following conditions:

   * used as Standard of Care outside ICU setting
   * could be removed for study drug administration (Note: oxygen flow at 2 L/min could be provided)

Ages: 28 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ablynx Clinical Department, Study Director — Ablynx, a Sanofi company
Locations (74):
- Belgium (5):
  - Investigator site 2, Brussels
  - Investigator site, Brussels
  - Investigator Site, Edegem
  - Investigator Site, Leuven
  - Investigator site, Roeselare
- Bulgaria (5):
  - Investigator Site, Kozloduy
  - Investigator Site, Plovdiv
  - Investigator Site, Rousse
  - Investigator Site, Sofia
  - Investigator Site, Stara Zagora
- Chile (2):
  - Investigator Site, Santiago
  - Investigator site, Valdivia
- Colombia (4):
  - Investigator site, Cali
  - Investigator Site, Floridablanca
  - Investigator Site 1, Medellín
  - Investigator site 2, Medellín
- Croatia (8):
  - Investigator site, Čakovec
  - Investigator site, Osijek
  - Investigator site, Slavonski Brod
  - Investigator site, Varaždin
  - Investigator site 1, Zagreb
  - Investigator site 2, Zagreb
  - Investigator site 3, Zagreb
  - Investigator site 4, Zagreb
- Investigator site, Hradec Králové, Czechia
- Investigator Site, Tartu, Estonia
- Germany (4):
  - Investigator site, Bochum
  - Investigator site, Dresden
  - Investigator Site, Sankt Augustin
  - Investigator Site, Wuppertal
- Hungary (9):
  - Investigator Site, Balassagyarmat
  - Investigator site 1, Budapest
  - Investigator Site 2, Budapest
  - Investigator Site 3, Budapest
  - Investigator Site 4, Budapest
  - Investigator site, Debrecen
  - Investigator Site, Szeged
  - Investigator site, Székesfehérvár
  - Investigator Site, Veszprém
- Israel (3):
  - Investigator site, Beersheba
  - Investigator site, Haifa
  - Investigator site, Petah Tikva
- Latvia (2):
  - Investigator Site, Daugavpils
  - Investigator Site, Riga
- Malaysia (4):
  - Investigator site, George Town
  - Investigator Site, Kuala Lumpur
  - Investigator Site, Seremban
  - Investigator Site, Sibu
- Philippines (4):
  - Investigator Site, Alabang
  - Investigator site, Manila
  - Investigator Site 1, Quezon City
  - Investigator Site 2, Quezon City
- Poland (2):
  - Investigator site, Lublin
  - Investigator site, Trzebnica
- Slovakia (4):
  - Investigator site, Banská Bystrica
  - Investigator site, Bratislava
  - Investigator site, Košice
  - Investigator Site, Poprad
- Spain (11):
  - Investigator Site 1, Barcelona
  - Investigator Site 2, Barcelona
  - Investigator Site 3, Barcelona
  - Investigator Site, Bilbao
  - Investigator Site, El Palmar
  - Investigator site 1, Madrid
  - Investigator Site 2, Madrid
  - Investigator Site, Málaga
  - Investigator site, Santiago de Compostela
  - Investigator site, Seville
  - Investigator Site, Valencia
- Thailand (5):
  - Investigator Site 1, Bangkok
  - Investigator site 2, Bangkok
  - Investigator Site, Chiang Mai
  - Investigator site, Hat Yai
  - Investigator Site, Khon Kaen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 301 subjects were screened.180 subjects were randomized to receive ALX-0171 3.0 mg/kg, ALX-0171 6.0 mg/kg, ALX-0171 9.0 mg/kg or placebo, yielding an overall allocation ratio of 3:1 active to placebo.
Groups:
- ALX-0171 9.0mg/kg: Inhalation of ALX-0171 9.0 mg/kg once daily for 3 consecutive days
Period: Overall Study
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Started (Intent-to-treat (ITT) Population: The ITT population consisted of all randomized subjects.) | 44 | 46 | 45 | 45
Included in the mITT Population (modified ITT (mITT): All randomized subjects who received at least 1 study drug administration.) | 42 | 45 | 43 | 45
Included in the Safety Population (Safety: All subjects who received at least 1 study drug administration, as treated.) | 40 | 45 | 44 (Includes a subject that was randomized to placebo but received a dose of ALX-0171 6.0 mg/kg) | 46 (Includes a subject that was randomized to placebo but received a dose of ALX-0171 9.0 mg/kg)
Completed | 40 | 44 | 43 | 44
Not Completed | 4 | 2 | 2 | 1
Not completed — Parent/guardian withdrew consent | 2 | 1 | 1 | 1
Not completed — Randomized but received no study drug | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Subject left country after Day14 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg | Total
Number analyzed (Participants) | 42 | 45 | 43 | 45 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 45 | 43 | 45 | 175
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] — The age reported is the age at the time of informed consent signing. Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  months | 6.964 (6.0668) | 6.933 (5.8827) | 6.657 (6.2605) | 7.022 (5.6884) | 6.896 (5.9234)
Age, Customized [Count of Participants; unit: Participants] — Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  Participants
    Age categories: < 6 months | 24 | 23 | 27 | 25 | 99
    Age categories: ≥ 6 months and < 12 months | 8 | 13 | 7 | 12 | 40
    Age categories: ≥ 12 months | 10 | 9 | 9 | 8 | 36
Age, Customized [Mean (Standard Deviation); unit: Weeks] — Age, Customized; Gestational Age Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  Weeks
    Gestational Age | 38.5 (1.78) | 38.6 (1.99) | 38.6 (1.62) | 38.3 (1.54) | 38.5 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  Participants
    Female | 24 | 15 | 19 | 17 | 75
    Male | 18 | 30 | 24 | 28 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  Participants
    Hispanic or Latino | 4 | 4 | 5 | 5 | 18
    Not Hispanic or Latino | 38 | 41 | 38 | 40 | 157
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  Participants
    Race: Asian | 7 | 7 | 3 | 10 | 27
    Race: Black or African American | 0 | 0 | 1 | 0 | 1
    Race: Multiple | 0 | 0 | 2 | 0 | 2
    Race: Other | 0 | 0 | 1 | 3 | 4
    Race: White | 35 | 38 | 36 | 32 | 141
Region of Enrollment [Count of Participants; unit: Participants] — Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  Participants
    Belgium | 2 | 3 | 3 | 1 | 9
    Bulgaria | 7 | 8 | 6 | 11 | 32
    Chile | 0 | 0 | 0 | 4 | 4
    Colombia | 0 | 0 | 1 | 0 | 1
    Croatia | 6 | 6 | 8 | 3 | 23
    Germany | 1 | 0 | 3 | 2 | 6
    Hungary | 7 | 6 | 8 | 4 | 25
    Israel | 0 | 2 | 1 | 1 | 4
    Latvia | 2 | 1 | 2 | 5 | 10
    Malaysia | 4 | 4 | 3 | 3 | 14
    Philippines | 1 | 1 | 0 | 3 | 5
    Poland | 5 | 5 | 3 | 0 | 13
    Slovakia | 0 | 0 | 2 | 2 | 4
    Spain | 5 | 7 | 2 | 1 | 15
    Thailand | 2 | 2 | 1 | 5 | 10
Number of days between symtpom onset and the first dose of study drug [Mean (Standard Deviation); unit: days] — Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  days | 3.16 (1.207) | 3.34 (1.144) | 3.23 (0.845) | 3.25 (1.149) | 3.25 (1.088)
Global Severity Score (GSS) [Mean (Standard Deviation); unit: score on a scale] — The GSS is a composite score based on the ReSVinet Scale (Justicia-Grande et al., 2016) that allowed for objective categorization of infants with respiratory infections based on seven different items (i.e., feeding intolerance, medical intervention, respiratory difficulty, respiratory frequency, apnea, general condition, and fever). The sum of the sub-item scores provides the GSS total score (range: 0-20). Higher score indicates more severe disease. Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  score on a scale | 9.1 (2.44) | 9.2 (2.00) | 9.3 (2.09) | 9.4 (2.41) | 9.2 (2.23)
Respiratory Distress Instrument (RDAI) [Mean (Standard Deviation); unit: score on a scale] — The RDAI instrument is a 17-point scoring system based on wheezing and retraction. The sum of the subscores provides the RDAI total score, with total range 0 to 17. Higher scores indicating more severe disease. Population: modified Intent-to-Treat Population (mITT): All randomized subjects who received at least 1 study drug administration. In this population, the subjects were classified as randomized (i.e.,using the treatment to which the subject was randomized).
  score on a scale | 8.5 (3.74) | 8.41 (4.07) | 8.74 (3.19) | 8.11 (3.80) | 8.44 (3.693)
Height [Mean (Standard Deviation); unit: centimetres] | 65.84 (9.997) | 65.71 (10.210) | 65.25 (10.190) | 66.55 (9.580) | 65.85 (9.915)
Weight [Mean (Standard Deviation); unit: kilograms] | 7.065 (2.4193) | 7.188 (2.2278) | 6.988 (2.4084) | 7.020 (2.2474) | 7.066 (2.3059)
Weight category [Count of Participants; unit: Participants]
  ≥ 3.0 kg and < 4.0 kg | 1 | 2 | 0 | 2 | 5
  ≥ 4.0 kg and < 5.0 kg | 8 | 6 | 13 | 7 | 34
  ≥ 5.0 kg and < 7.0 kg | 15 | 15 | 11 | 14 | 55
  ≥ 7.0 kg and < 10.0 kg | 11 | 17 | 12 | 19 | 59
  ≥ 10.0 kg and < 12.0 kg | 6 | 4 | 7 | 1 | 18
  ≥ 12.0 kg and < 15.0 kg | 1 | 1 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time for Viral Load to Drop Below Assay Quantification Limit (BQL) (Plaque Assay Analysis)
Description: The primary endpoint for this trial was the time needed for the viral load to drop below the quantification limit (time-to-BQL) of the plaque assay in nasal mid-turbinate swab specimens. Time-to-BQL was defined as the time from the first study drug administration to the first occurrence of a value below the quantification limit (BQL), provided the next measured value was also below the limit of quantification. The time to BQL for subjects with missing data and/or who did not reach BQL during the trial were censored at the last non-missing viral load assessment. The primary endpoint was analysed using logrank test to compare time-to-BQL between each of the ALX-0171 treatment groups and the combined placebo group. The tests were performed in a sequential way to preserve the family-wise error rate at 0.05. The comparisons were performed in the following order: ALX-0171 9 mg/kg vs Placebo, followed by ALX-0171 6mg/kg vs Placebo, ALX-0171 3mg/kg vs Placebo.
Time Frame: Overall Study Period (i.e., approximately 28 days)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 42 | 45 | 43 | 45
hours | 46.1 [29.33 to 94.42] | 14.2 [5.17 to 26.28] | 5.1 [4.78 to 24.72] | 5.1 [4.97 to 5.17]
Statistical Analysis 1: Comparison: Placebo vs ALX-0171 9.0mg/kg; The primary endpoint was analysed using log-rank test to compare time-to-BQL between each of the ALX-0171 treatment groups and the combined placebo group. The tests were performed in a sequential way to preserve the family-wise error rate at 0.05; Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 2: Comparison: Placebo vs ALX-0171 6.0 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Log Rank
Statistical Analysis 3: Comparison: Placebo vs ALX-0171 3.0 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Log Rank

2. Secondary Outcome: Change From Baseline in Global Severity Score on Day 2 (5 Hours Post-dose)
Description: A formal comparison for change from Baseline in GSS to Day 2, 5 hours post-dose was performed using a contrast analysis on a longitudinal mixed model with random factor subject and fixed effects baseline value, treatment group and timepoint, including the treatment-by-timepoint interaction term. All data up to and including Day 3 were used in the longitudinal mixed model. The Kenward-Roger approximation of degrees of freedom was used. The model was fitted using an unstructured variance-covariance matrix.
  The individual pair-wise comparisons were reported (comparison in least square [LS] means for 9.0 mg/kg versus placebo; 6.0mg/kg versus placebo; 3.0 mg/kg versus placebo).
  Evolution over time in Global Severity Score. The maximum total score is 20 (minimum:0 to manimum:20); higher score indicates more severe disease.
Time Frame: from Baseline untill Day 2 (5 hours post-dose)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 42 | 45 | 43 | 45
score on a scale | -3.6392 (0.4160) | -3.8548 (0.4103) | -4.1296 (0.4129) | -4.2844 (0.4099)
Statistical Analysis 1: Comparison: Placebo vs ALX-0171 9.0mg/kg; A comparison for change from Baseline in GSS to Day 2, 5 hours post-dose was performed using a contrast analysis on a longitudinal mixed model with random factor subject and fixed effects baseline value, treatment group and timepoint, including the treatment-by-timepoint interaction term. All data up to + including Day 3 were used in the longitudinal mixed model. The Kenward-Roger approximation of degrees of freedom was used.The model was fitted using an unstructured variance-covariance matrix; Test type: Superiority; p = 0.271, Mixed Models Analysis; Mean Difference (Net) = -0.6452, Standard Error of Mean 0.5843
Statistical Analysis 2: Comparison: Placebo vs ALX-0171 6.0 mg/kg; Test type: Superiority; p = 0.404, Mixed Models Analysis; Difference in LS means = -0.4904, Standard Error of Mean 0.5862
Statistical Analysis 3: Comparison: Placebo vs ALX-0171 3.0 mg/kg; Test type: Superiority; p = 0.713, Mixed Models Analysis; Difference in LS means = -0.2156, Standard Error of Mean 0.5842

3. Secondary Outcome: Time-to-Clinical Response
Description: The time-to-clinical response was defined as the time between the first study drug administration and the time of achieving adequate oxygen saturation (defined as SpO2 > 92% over a period of at least 4 hours) and adequate oral feeding (which is sufficient to maintain sufficient hydration, in the judgment of the Investigator).
Time Frame: Overall Study Period (i.e., approximately 28 days)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 42 | 45 | 43 | 45
hours
  Time-to-Clinical Response | 47.9 [29.17 to 64.08] | 44.1 [28.33 to 51.20] | 27.9 [21.08 to 43.68] | 46.3 [38.00 to 50.38]
  Time-to-adequate oral feeding | 43.7 [22.50 to 47.58] | 44.0 [25.92 to 52.00] | 17.6 [6.50 to 25.85] | 23.8 [17.17 to 38.00]
  Time-to-adequate oxygen saturation | 53.4 [28.70 to 71.78] | 38.5 [24.75 to 61.93] | 29.5 [20.75 to 47.43] | 46.5 [42.15 to 48.25]

4. Secondary Outcome: Time-to-BQL (RT-qPCR)
Description: As secondary endpoint, the time-to-BQL using RT-qPCR was summarized using Kaplan Meier (KM) estimates. No p-values were calculated. For RSV load by RT-qPCR, the lower limit of quantification (LLOQ) was 2.4 log10 copies/mL.
  The upper limit confidence interval (CI) could not be calculated; Values of the 25 percentile are reported here.
Time Frame: Overall Study Period (i.e., approximately 28 days)
Population: The modified ITT (mITT) population consisted of all randomized subjects who received at least 1 administration of study drug. When using this population, the subjects were classified as randomized (i.e., using the treatment to which the subject was randomized).
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 42 | 45 | 43 | 45
hours | 26.7 [5.0 to 49.92] | 26.8 [5.17 to 44.62] | 28.9 [18.25 to 49.25] | 6.3 [4.97 to 25.25]

5. Secondary Outcome: Time-to-undetectable Viral Load (Plaque Assay Analysis)
Description: The time-to-undetectability (hours), defined as the time from the first study drug administration to the first occurrence of viral titer below the lower limit of quantification (LLOQ), and target not detected provided the next measured value was also below the quantification limit and undetected, were summarized using KM estimates, based on the plaque assay. The time-to-event for subjects with missing data and/or subjects who did not reach undetectability during the trial were censored at the last non-missing viral load assessment. For RSV load by plaque assay the LLOQ was 1.7 log10 pfu/mL.
Time Frame: Overall Study Period (i.e., approximately 28 days)
Population: RSV-Infected Population: A central RSV test was used for defining the RSV-Infected population. The RSV-Infected population consisted of all randomized subjects with RSV infection, as confirmed by RT-qPCR (hVIVO quantitative PCR assay) on Day 1 (pre- or post-dose), who received at least 1 administration of study drug.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 35 | 40 | 40 | 38
hours | 95.9 [47.23 to 121.82] | 26.3 [20.25 to 28.92] | 21.0 [4.88 to 28.25] | 5.1 [5.00 to 5.87]

6. Secondary Outcome: Viral Load Changes From Baseline (Plaque Assay Analysis)
Description: Change from Baseline in RSV Load measured by Plaque Assay (RSV Infected Population)
Time Frame: From Baseline until Day 14 (Follow-up) (Baseline; Day 1, 5 hours post-dose; Day 3, 2 hours post-dose; and Follow-up reported)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: log10 pfu/mL
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 35 | 40 | 40 | 38
log10 pfu/mL
  Baseline | 3.494 (0.2396) | 3.312 (0.2165) | 3.135 (0.2430) | 2.385 (0.2526)
  Day 1, 5 hours post-dose | -0.270 (0.1607) | -2.173 (0.2123) | -2.189 (0.2676) | -1.535 (0.2526)
  Day 3, 2 hours post-dose | -1.936 (0.2317) | -2.396 (0.2234) | -2.134 (0.2525) | -1.516 (0.2558)
  Follow-up | -2.368 (0.2946) | -2.431 (0.2202) | -2.279 (0.2576) | -1.416 (0.2821)

7. Secondary Outcome: Viral Load Changes From Baseline (RT-qPCR Analysis)
Description: Change from Baseline in RSV Load measured by RT-qPCR (RSV Infected Population)
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 35 | 40 | 40 | 38
log10 copies/mL
  Baseline | 5.236 (0.2827) | 4.966 (0.2095) | 5.232 (0.1899) | 4.525 (0.2937)
  Day 1, 5 hours post-dose | -0.221 (0.1601) | -0.544 (0.1286) | -0.241 (0.2031) | -0.449 (0.1883)
  Day 3, 2 hours post-dose | -2.156 (0.2454) | -2.589 (0.2138) | -2.310 (0.2797) | -2.025 (0.2840)
  Follow-up | -3.413 (0.3715) | -3.665 (0.2203) | -3.972 (0.2032) | -3.033 (0.3252)

8. Secondary Outcome: Viral Load Time-weighted Average Changes From Baseline (Plaque Assay Analysis)
Description: The time-weighted average change from baseline to Day x was defined as (AUCx - x* viral load at baseline) /x, where AUCx denotes the AUC between baseline and Day x. For subjects who only had data up to Day t (t<x), the endpoint was defined as (AUCt - t*viral load at baseline) / t.
Time Frame: From Baseline until Day 14 (Follow-up) (Baseline, Day 3, and Follow-up reported)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: log10 pfu/mL
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 35 | 40 | 40 | 38
log10 pfu/mL
  Baseline | 3.494 (0.2396) | 3.312 (0.2165) | 3.135 (0.2430) | 2.385 (0.2526)
  Day 3 | -1.014 (0.1540) | -1.924 (0.1659) | -1.804 (0.2098) | -1.330 (0.2434)
  Follow-Up | -2.096 (0.2443) | -2.295 (0.2116) | -2.028 (0.2217) | -1.419 (0.2488)

9. Secondary Outcome: Viral Load Time-weighted Average Changes From Baseline (RT-qPCR Analysis)
Description: as for outcome 8
Time Frame: From Baseline until Day 14 (Follow-up) (Baseline, Day 3, and Follow-up reported)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 35 | 40 | 40 | 38
log10 copies/mL
  Baseline | 5.236 (0.2827) | 4.966 (0.2095) | 5.232 (0.1899) | 4.525 (0.2937)
  Day 3 | -0.933 (0.1421) | -1.209 (0.1301) | -1.113 (0.1932) | -0.842 (0.1842)
  Follow-up | -2.684 (0.2263) | -2.828 (0.2099) | -2.756 (0.1831) | -2.292 (0.2581)

10. Secondary Outcome: Immunogenicity; Number of Subjects With Treatment-emergent Anti-drug Antibodies
Description: The number of subjects with treatment-emergent (TE) anti-drug antibodies (ADA; TE ADA) based on ADA assay by treatment group for the Safety Population. Blood samples for immunogenicity assessments were collected at Baseline and on Day 14.
  Immunogenicity data were analyzed using the Safety Population. This population differs from the ITT and mITT Populations as 2 subjects who were originally randomized to placebo, received active treatment once; one subject received ALX-0171 6.0 mg/kg and one subject ALX-0171 9.0 mg/kg.
Time Frame: Overall Study Period (i.e., approximately 28 days)
Population: The Safety Population consisted of all subjects who received at least 1 administration of study drug. When using this population, the subjects were classified as treated (i.e., using the treatment that the subject actually received). Number of subjects with non-missing ADA results were: placebo:39; ALX-0171 3.0mg/kg:45; 6.0mg/kg:44; 9.0mg/kg:46.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 39 | 45 | 44 | 46
Participants
  Total TE ADA Positive | 10 | 15 | 16 | 15
  Total TE ADA Negative | 16 | 17 | 14 | 13
  TE ADA Equivocal | 12 | 12 | 13 | 14
  TE ADA Inconclusive | 1 | 1 | 1 | 4

11. Secondary Outcome: Immunogenicity; Number of Subjects With Treatment-emergent Neutralizing Antibodies
Description: Number of subjects with treatment-emergent neutralizing antibodies (TE NAb) as detected with the competitive ligand binding NAb assay. Blood samples for immunogenicity assessments were collected at Baseline and on Day 14.
  Immunogenicity data were analyzed using the Safety Population. This population differs from the ITT and mITT Populations as 2 subjects who were originally randomized to placebo, received active treatment once; one subject received ALX-0171 6.0 mg/kg and one subject ALX-0171 9.0 mg/kg.
Time Frame: Overall Study Period (i.e., approximately 28 days)
Population: The Safety Population consisted of all subjects who received at least 1 administration of study drug. When using this population, the subjects were classified as treated (i.e., using the treatment that the subject actually received).Number of subjects with non-missing NAb results were: placebo:39; ALX-0171 3.0mg/kg:45; 6.0mg/kg:44; 9.0mg/kg:46.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
Number analyzed (Participants) | 39 | 45 | 44 | 46
Participants
  Post-dose Positive | 2 | 11 | 18 | 12
  Post-dose Negative | 36 | 33 | 26 | 31
  Post-dose Missing | 1 | 1 | 0 | 3

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were reported from first study drug intake to the end of study visit (Day 28) or withdrawal visit.
Description: A treatment-emergent AE (TEAE) was defined as any AE starting or worsening in severity (for preexisting conditions) from the start of study drug administration, until completion of the subject's last visit.
  Adverse event data were analyzed using the Safety Population. This population differs from the ITT and mITT Populations as 2 subjects who were originally randomized to placebo, received active treatment once; one subject received ALX-0171 6.0 mg/kg and one subject ALX-0171 9.0 mg/kg.
Arm/Group | Placebo | ALX-0171 3.0 mg/kg | ALX-0171 6.0 mg/kg | ALX-0171 9.0mg/kg
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/45 | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 5/40 | 4/45 | 3/44 | 3/46
Other Adverse Events (participants affected / at risk) | 17/40 | 16/45 | 16/44 | 10/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | ALX-0171 3.0 mg/kg (N=45) | ALX-0171 6.0 mg/kg (N=44) | ALX-0171 9.0mg/kg (N=46)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | ALX-0171 3.0 mg/kg (N=45) | ALX-0171 6.0 mg/kg (N=44) | ALX-0171 9.0mg/kg (N=46)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (4) | 2 (2)
Conjuctivitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Otitis media (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02979431/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT02979431/SAP_001.pdf